CLINICAL TRIAL: NCT03932006
Title: A Multicenter，Double-Blind and Randomized Controlled Trial of Fengshigutong Capsule in the Treatment of Ankylosing Spondylitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Division of Rheumatology of Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: [2015]2-159
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; Fengshigutong Capsule; imrecoxib
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Imrecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fengshigutong Capsule plus Imrecoxib (Experimental): Fengshigutong Capsule 1.2g twice a day,Imrecoxib 0.1g twice a day,orally
  Interventions: Drug: Fengshigutong Capsule plus Imrecoxib
- Fengshigutong Capsule (Experimental): Fengshigutong Capsule 1.2g twice a day,orally
  Interventions: Drug: Fengshigutong Capsule
- Imrecoxib (Active Comparator): Imrecoxib 0.1g twice a day,orally
  Interventions: Drug: Imrecoxib

INTERVENTIONS:
Drug: Fengshigutong Capsule plus Imrecoxib — Fengshigutong Capsule 1.2g twice a day,Imrecoxib 0.1g twice a day,orally
  Arms: Fengshigutong Capsule plus Imrecoxib
Drug: Fengshigutong Capsule — Fengshigutong Capsule 1.2g twice a day,orally
  Arms: Fengshigutong Capsule
Drug: Imrecoxib — Imrecoxib 0.1g twice a day,orally
  Arms: Imrecoxib

SUMMARY:
This is a randomized, double-blind, multicentral clinical trial to investigate the efficacy and safety of Fengshigutong Capsule in the treatment of active ankylosing spondylitis(AS). The primary purpose is to assess the different maintaining treatment programme in AS patients with controlled inflammation by Imrecoxib. The trial will include 180 patients who will be divided into three group: Fengshigutong Capsule plus Imrecoxib group, Imrecoxib group and Fengshigutong Capsule group. Patients will complete the 4-week therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years
* Meet 1984 modified New York criteria for AS
* The Bath AS Disease Activity Index (BASDAI) ≥4 on a 0-10-cm visual analog scale or the Ankylosing Spondylitis Disease Activity Score using the C-reactive protein level (ASDAS-CRP) ≥1.3
* NSAIDs washout period of at least 7 days prior to randomization
* DMARDs washout period of at least 4 weeks prior to randomization
* Corticosteroids washout period of at least 2 weeks prior to randomization
* Biological agents washout period of at least 3 months prior to randomization.

Exclusion Criteria:

* Peptic ulcer
* Unstable cardiac diseases
* Hematologic disorders
* Psychosis
* Malignancy
* Multiple sclerosis
* severe COPD
* fibromyalgia and other rheumatic disease
* Corticosteroids were injected into the articular cavity within 3 months
* Chinese medicine was taken within 28 days
* Pregnant and lactating women
* Alcohol and drug abuse
* Spinal cord compression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06-30 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
the proportions of patients reaching Assessment in Ankylosing Spondylitis 20% | 4 week
  ASAS20 was defined as an improvement of ≥20% and absolute improvement of ≥1 unit (0-10-cm VAS) from baseline in ≥3 of the following 4 domains (and absence of deterioration in any domain): patient's global assessment of disease activity (PTGA), pain assessment (mean of total and nocturnal pain scores), Bath Ankylosing Spondylitis Functional Index (BASFI), and clinical inflammation (mean of 2 morning stiffness-related scores on the BASDAI)

SECONDARY OUTCOMES:
the proportions of patients reaching Assessment in Ankylosing Spondylitis 50% | 4 week
  defined as 20% improvement in 5 of the following 6 domains: PTGA, pain assessment, BASFI, clinical inflammation, spinal mobility, and C-reactive protein (CRP)
ASAS20 response | 4 week
  ASAS20 was defined as an improvement of ≥20% and absolute improvement of ≥1 unit (0-10-cm VAS) from baseline in ≥3 of the following 4 domains (and absence of deterioration in any domain): patient's global assessment of disease activity (PTGA), pain assessment (mean of total and nocturnal pain scores), Bath Ankylosing Spondylitis Functional Index (BASFI), and clinical inflammation (mean of 2 morning stiffness-related scores on the BASDAI)
ASAS5/6 response | 4 week
  defined as 20% improvement in 5 of the following 6 domains: PTGA, pain assessment, BASFI, clinical inflammation, spinal mobility, and C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, Prof, Study Director — Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China